CLINICAL TRIAL: NCT01065350
Title: A Comparison of Ketofol (Ketamine and Propofol Admixture) vs. Propofol as Induction Agents on Hemodynamic Parameters
Brief Title: A Comparison of Ketofol (Ketamine and Propofol Admixture) Versus Propofol as Induction Agents on Hemodynamic Parameters
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Principal Investigator, Nathan J. Smischney, PI, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 22063
Record Dates: First submitted 2010-02-07; First posted 2010-02-09 (Estimated); Results first posted 2013-05-03 (Estimated); Last update posted 2013-05-03 (Estimated); Status verified 2013-03

CONDITIONS: Blood Pressure
Keywords: ketofol; hemodynamics; propofol; anesthesia
MeSH Terms: interventions — Propofol; Ketamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Propofol (Active Comparator): As part of the induction, patients will be given 2 milligrams of propofol per kilogram (mg/kg) of body weight. The clinician will receive a 20 milliliter (mL) syringe of propofol. If the dose, 2 mg/kg, does not add up to a total of 20 mL, normal saline will be added to make up for the 20 mL.
  Interventions: Drug: Propofol
- Ketofol (Experimental): As part of the induction, patients will be given 20 mL syringe of an admixture called "ketofol," which combines ketamine and propofol in one syringe. The dose is weight-based such that ketamine will represent 0.75 mg/kg of the dose and propofol, 1.5 mg/kg of the dose.
  Interventions: Drug: Ketamine

INTERVENTIONS:
Drug: Propofol — As part of the induction, subjects will be given 2 milligrams per kilogram of body weight (mg/kg) of propofol. The clinician will receive a 20 milliliter (mL) syringe of propofol. If the dose, 2 mg/kg, does not add up to a total of 20 mL, normal saline will be added to make up for the 20 mL. The clinician and observer will be blinded to the medication and doses being administered during induction given that both syringes, syringes in the propofol and ketofol groups, will look identical (will both appear to be propofol only). The propofol group will also be given an additional 10 mL syringe of propofol due to any patient responding to stimulus after induction. The 10 mL syringe represents 1 mg/kg of propofol. If patient receives both the 20 and 10ml syringe, he or she will receive a total of 3mg/kg of propofol.
  Other Names: Diprivan
  Arms: Propofol
Drug: Ketamine — As part of the induction, patients will be given 20ml syringe of ketofol which is weight based such that ketamine will represent 0.75mg/kg of the dose and propofol, 1.5mg/kg. The clinician and observer will be blinded to the medication and doses being administered during induction given that both 20ml syringes (propofol group and ketofol group) will look identical (will both appear to be propofol only). Additional 10ml syringe will be given due to any patient responding to stimulus after induction. The 10ml syringe will represent 0.25mg/kg of ketamine and 0.5mg/kg of propofol. If the patient receives both the 20 and 10ml rescue syringe, he or she will receive a total of 1mg/kg of ketamine and 2mg/kg of propofol.
  Other Names: Ketalar
  Arms: Ketofol

SUMMARY:
This is a pilot study to compare the hemodynamic changes that occur during induction with a novel drug combination known as ketofol (propofol and ketamine admixture with that of propofol alone (prototypic anesthesia induction agent). Propofol and ketamine are widely used as induction agents and their effects on patient hemodynamics are well known. Some of these drug-induced hemodynamic changes are undesirable and lead to deleterious effects on patient hemodynamics. We seek to investigate the hemodynamic changes associated with a novel drug combination known as ketofol (ketamine/propofol admixture) during induction and compare them to propofol. If we determine that the changes produced by ketofol are favorable compared with propofol, we then will seek to test its use in the trauma setting in a subsequent randomized controlled trial.

DETAILED DESCRIPTION:
This is a pilot study to compare the hemodynamic changes that occur during induction with a novel drug combination known as ketofol with that of propofol. Propofol and ketamine are widely used as induction agents and their effects on patient hemodynamics are well known. Many of these drug-induced changes are undesirable and when used alone sometimes lead to hemodynamic effects on opposite ends of the spectrum, ie. hypotension (propofol) and hypertension (ketamine). We will investigate the hemodynamic changes associated with this drug combination referred to as "ketofol" (ketamine/propofol admixture) during induction compared with propofol as the gold standard induction agent used widely in anesthetic practice. If we validate that the changes produced by the ketofol admixture are favorable, we will then test its use in a wider setting of patient populations including emergency department intubations and the trauma setting.

Background: Propofol is a non-opioid, non-barbiturate, sedative-hypnotic agent with rapid onset and short duration of action. It possesses many favorable effects such as an antiemetic effect and reliably produces sedation and amnesia (Felfernig Jour of Royal Naval Medical Service, '06; White International Anesth Clinics, '88; Willman Ann of Emer Med, '07). However, there are several undesirable side effects such as cardiovascular and respiratory depression. In addition, Propofol as a sole agent has no analgesic properties. These drug-induced side effects have led to alternative drugs being used with the hopes of a more favorable side effect profile. Ketamine is an example of one such drug. Ketamine is a phencyclidine derivative commonly classified as a dissociative sedative with fairly rapid onset and short duration of action (Felfernig Jour of Royal Naval Medical Service, '06; White International Anesth Clinics, '88; Willman Ann of Emer Med, '07). It causes little or no respiratory and cardiovascular depression and unlike propofol, has pain relieving properties. Ketamine as a single induction agent, however, is limited by emergence phenomena including postoperative dreaming and hallucinations, however these are attenuated by the administration of benzodiazepines. Also ketamine in induction doses 1-4.5 mg/kg can have some undesirable effects on hemodynamics (opposite of propofol) in certain patient populations including ischemic heart disease (IHD), and patients with increases in intracranial hypertension and intracranial pressure (ICP). Effectiveness of the two agents in combination has been recently demonstrated and this new combination could allow a novel induction agent with favorable effects on hemodynamics (Felfernig Jour of Royal Naval Medical Service, '06; Hui Jour of Amer Soc of Anesth, '95; Willman Ann of Emer Med, '07). To date, this combination known as ketofol has been used most extensively for procedural sedation in the Emergency Department but has not yet been standardized as an induction agent. We are obtaining funding for a pilot study to validate the use of ketofol as an induction agent.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) physical status I and II who are to undergo elective general, urologic, orthopedic, plastic, or gynecologic surgery.

Exclusion Criteria:

* patients with age less than 18 yr or over 60 yr,
* emergency surgery,
* patients undergoing neurosurgical procedures,
* any procedure with adjunctive analgesia,
* any patient on chronic opiate use,
* females who are known to be pregnant,
* patients who had ingested psychotropic or sedative medication within one month of investigation,
* patients with personality disorders,
* weight greater than 20% of ideal, and
* any known contraindications to ketamine or propofol.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 85 (Actual)
Dates: Start 2010-12; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nathan J Smischney, MD, Principal Investigator — Mayo Clinic; Matthew Koff, MD, Study Director — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire, United States

REFERENCES:
- [Result] Smischney NJ, Beach ML, Loftus RW, Dodds TM, Koff MD. Ketamine/propofol admixture (ketofol) is associated with improved hemodynamics as an induction agent: a randomized, controlled trial. J Trauma Acute Care Surg. 2012 Jul;73(1):94-101. doi: 10.1097/TA.0b013e318250cdb8. PMID 22743378

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients requiring surgical procedures with general anesthesia were recruited and enrolled at Dartmouth-Hitchcock Medical Center in Lebanon, New Hampshire from December 2010 to March 2011.
Period: Overall Study
Arm/Group | Propofol | Ketofol
Started | 43 | 42
Completed | 43 | 41
Not Completed | 0 | 1
Not completed — Received incorrect drug allocation | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Ketofol: As part of the induction, patients will be given 20 mL syringe of an admixture called "ketofol," which combines ketamine and propofol in one syringe. The dose is weight-based such that ketamine will represent 0.75 mg/kg of the dose and propofol, 1.5 mg/kg of the dose. One subject in the ketofol group was excluded from analysis due to incorrect study drug assignment and outside the protocol-specified dose.
- Total: Total of all reporting groups
Arm/Group | Propofol | Ketofol | Total
Number analyzed (Participants) | 43 | 41 | 84
Age Continuous [Mean (Standard Deviation); unit: years] | 43 (11) | 42 (12) | 42.68 (11.51)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 27 | 55
  Male | 15 | 14 | 29
Region of Enrollment [Number; unit: participants]
  United States | 43 | 41 | 84
Body Weight [Mean (Standard Deviation); unit: kilograms] | 69.2 (11.7) | 68.9 (11.2) | 68.97 (11.41)
Body Height [Mean (Standard Deviation); unit: centimeters] | 169.9 (9.1) | 168.9 (9.2) | 169.40 (9.03)
Systolic Blood Pressure [Mean (Standard Deviation); unit: millimeters of mercury (mm Hg)] — Mean pre-operative systolic blood pressure
  millimeters of mercury (mm Hg) | 125 (17) | 122 (15) | 124.19 (16.41)
Diastolic Blood Pressure [Mean (Standard Deviation); unit: millimeters of mercury (mm Hg)] — Mean pre-operative diastolic blood pressure
  millimeters of mercury (mm Hg) | 76 (12) | 76 (10) | 76 (11)
Heart Rate [Mean (Standard Deviation); unit: beats per minute] — Mean pre-operative heart rate
  beats per minute | 72 (16) | 73 (14) | 73 (15)
American Society of Anesthesiology (ASA) Physical Status [Number; unit: Participants] — ASA Physical Status 1 - A normal healthy patient
  ASA Physical Status 2 - A patient with mild systemic disease
  Participants
    ASA Status 1 | 21 | 14 | 35
    ASA Status 2 | 22 | 27 | 49

OUTCOME MEASURES:

1. Primary Outcome: Percent of Subjects With a Greater Than 20% Decrease in Systolic Blood Pressure (SBP) Following Induction of General Anesthesia
Description: Blood pressure was recorded every minute for a total of 30 minutes after anesthesia was induced and readings were captured via a Non-Invasive Cardiac Output Monitor [NICOM], Cheetah Medical, Israel. The percentage of subjects experiencing decreases in SBP of greater than 20% during the specified time intervals is reported, as compared to the baseline systolic blood pressure reading. There are two numbers in a blood pressure reading, and they are expressed in millimeters of mercury (mm Hg). This tells how high in millimeters the pressure of your blood raises a column of mercury. The numbers usually are expressed in the form of a fraction; an example of a blood pressure reading is 120/80 mm Hg. The first, or top, number (120 in the example) is the systolic pressure. The systolic pressure is the measure of your blood pressure as the heart contracts and pumps blood.
Time Frame: Baseline, 5 minutes, 10 minutes, 30 minutes post induction
Population: 85 patients were enrolled (43 Propofol/42 Ketofol). However, one subject randomized to the ketofol group received the wrong study drug and in a larger dose than indicated in protocol. This subject was excluded from the analysis and baseline measures.
Measure: Number; unit: Percentage of subjects
Arm/Group | Propofol | Ketofol
Number analyzed (Participants) | 43 | 41
Percentage of subjects
  SBP baseline to 5 minutes | 48 [2.07 to 26.15] | 12
  SBP baseline to 10 minutes | 67 | 39
  SBP baseline to 30 minutes | 76 | 68
Statistical Analysis 1: Comparison: Propofol vs Ketofol; Systolic Blood Pressure (SBP) from baseline to 5 minutes post induction was compared between treatment groups; Test type: Superiority or Other; p < 0.001, Chi-squared — A p value of < 0.05 was considered to indicate statistical significance; Odds Ratio (OR) = 6.87, 95% CI 2-sided [2.07 to 26.15]
Statistical Analysis 2: Comparison: Propofol vs Ketofol; Systolic Blood Pressure (SBP) from baseline to 10 minutes post induction was compared between treatment groups; Test type: Superiority or Other; p < 0.01, Chi-squared — A p value of < 0.05 was considered to indicate statistical significance; Odds Ratio (OR) = 3.24, 95% CI 2-sided [1.21 to 8.75]
Statistical Analysis 3: Comparison: Propofol vs Ketofol; Systolic Blood Pressure (SBP) from baseline to 30 minutes post induction was compared between treatment groups; Test type: Superiority or Other; p = 0.39, Chi-squared — A p value of < 0.005 was considered to indicate statistical significance; Odds Ratio (OR) = 1.53, 95% CI 2-sided [0.52 to 4.55]

2. Secondary Outcome: Percent of Subjects With a Greater Than 20% Decrease in Diastolic Blood Pressure (DBP) Following Induction of General Anesthesia
Description: Blood pressure was recorded every minute for a total of 30 minutes after anesthesia was induced and readings were captured via a Non-Invasive Cardiac Output Monitor [NICOM], Cheetah Medical, Israel. The percentage of subjects experiencing decreases in DBP of greater than 20% during the specified time intervals is reported, as compared to the baseline DBP reading. The second or lower number of a blood pressure reading is the DBP and is the measure taken when your heart is at rest.
Time Frame: Baseline, 5 minutes, 10 minutes, 30 minutes post induction
Population: as for outcome 1
Measure: Number; unit: Percentage of subjects
Arm/Group | Propofol | Ketofol
Number analyzed (Participants) | 43 | 41
Percentage of subjects
  DBP baseline to 5 minutes | 48 | 17
  DBP baseline to 10 minutes | 62 | 41
  DBP baseline to 30 minutes | 90 | 78
Statistical Analysis 1: Comparison: Propofol vs Ketofol; Diastolic Blood Pressure (DBP) from baseline to 5 minutes post induction was compared between treatment groups; Test type: Superiority or Other; p < 0.01, Chi-squared — A p value of < 0.05 was considered to indicate statistical significance; Odds Ratio (OR) = 4.64, 95% CI 2-sided [1.54 to 14.92]
Statistical Analysis 2: Comparison: Propofol vs Ketofol; Diastolic Blood Pressure (DBP) from baseline to 10 minutes post induction was compared between treatment groups; Test type: Superiority or Other; p = 0.05, Chi-squared — A p value of < 0.05 was considered to indicate statistical significance; Odds Ratio (OR) = 2.38, 95% CI 2-sided [0.91 to 6.29]
Statistical Analysis 3: Comparison: Propofol vs Ketofol; Diastolic Blood Pressure (DBP) from baseline to 30 minutes post induction was compared between treatment groups; Test type: Superiority or Other; p = 0.11, Chi-squared — A p value of < 0.05 was considered to indicate statistical significance; Odds Ratio (OR) = 2.74, 95% CI 2-sided [0.68 to 13.19]

3. Secondary Outcome: Percent of Subjects With a Greater Than 20% Decrease in Mean Arterial Pressure (MAP) Following Induction of General Anesthesia
Description: MAP was recorded every minute for a total of 30 minutes after anesthesia was induced and readings were captured via a Non-Invasive Cardiac Output Monitor [NICOM], Cheetah Medical, Israel. The percentage of subjects experiencing decreases in MAP of greater than 20% during the specified time intervals is reported, as compared to the baseline MAP reading.
Time Frame: Baseline, 5 minutes, 10 minutes, 30 minutes post induction
Population: as for outcome 1
Measure: Number; unit: Percentage of subjects
Arm/Group | Propofol | Ketofol
Number analyzed (Participants) | 43 | 41
Percentage of subjects
  MAP baseline to 5 minutes | 44 | 10
  MAP baseline to 10 minutes | 60 | 35
  MAP baseline to 30 minutes | 83 | 75
Statistical Analysis 1: Comparison: Propofol vs Ketofol; Mean Arterial Pressure (MAP) from baseline to 5 minutes post induction was compared between treatment groups; Test type: Superiority or Other; p < 0.001, Chi-squared — A p value of < 0.05 was considered to indicate statistical significance; Odds Ratio (OR) = 7.12, 95% CI 2-sided [1.98 to 31.64]
Statistical Analysis 2: Comparison: Propofol vs Ketofol; Mean Arterial Pressure (MAP) from baseline to 10 minutes post induction was compared between treatment groups; Test type: Superiority or Other; p = 0.02, Chi-squared — A p value of < 0.05 was considered to indicate statistical significance; Odds Ratio (OR) = 2.84, 95% CI 2-sided [1.07 to 7.65]
Statistical Analysis 3: Comparison: Propofol vs Ketofol; Mean Arterial Pressure (MAP) from baseline to 30 minutes post induction was compared between treatment groups; Test type: Superiority or Other; p = 0.33, Chi-squared — A p value of < 0.05 was considered to indicate statistical significance; Odds Ratio (OR) = 1.71, 95% CI 2-sided [0.51 to 5.97]

4. Secondary Outcome: Average Change in Cardiac Output (CO)
Description: CO was recorded every minute for a total of 30 minutes after anesthesia was induced and readings were captured via a Non-Invasive Cardiac Output Monitor [NICOM], Cheetah Medical, Israel. The average change in CO as compared to baseline CO during the specified time intervals is reported.
  CO is defined as the quantity of blood ejected per minute by the heart into the systemic circulation. It is the product of the heart rate (HR) (beats per minute) times the stroke volume (SV) (milliliters of blood ejected during each contraction).
Time Frame: Baseline, 5 minutes, 10 minutes post induction
Population: The analysis population of 41/40 (vs. 43/41 at baseline) is due to the NICOM not functioning properly during certain aspects of the procedure and therefore, did not provide a number.
Measure: Mean (Standard Deviation); unit: Liters per minute
Arm/Group | Propofol | Ketofol
Number analyzed (Participants) | 41 | 40
Liters per minute
  5 minutes post induction | -0.8 (0.8) | -0.6 (0.6)
  10 minutes post induction | -1.0 (1.0) | -0.9 (0.8)
Statistical Analysis 1: Comparison: Propofol vs Ketofol; Average change in Cardiac Output (CO) from baseline to 5 minutes post induction was compared between treatment groups; Test type: Superiority or Other; p = 0.19, t-test, 2 sided; Mean Difference (Final Values) = 0.2, 95% CI 2-sided [-0.1 to 0.5]
Statistical Analysis 2: Comparison: Propofol vs Ketofol; Average change in Cardiac Output (CO) from baseline to 10 minutes post induction was compared between treatment groups; Test type: Superiority or Other; p = 0.6, t-test, 2 sided; Mean Difference (Final Values) = 0.1, 95% CI 2-sided [-0.3 to 0.5]

5. Secondary Outcome: Average Change in Cardiac Index (CI)
Description: CI was recorded every minute for a total of 30 minutes after anesthesia was induced and readings were captured via a Non-Invasive Cardiac Output Monitor [NICOM], Cheetah Medical, Israel. The average change in CI as compared to the baseline CI during the specified time intervals is reported.
  To determine CI, cardiac output is divided by the body surface area in order to account for body size.
Time Frame: Baseline, 5 minutes, 10 minutes post induction
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Liters per minute per m^2 of body area
Arm/Group | Propofol | Ketofol
Number analyzed (Participants) | 41 | 40
Liters per minute per m^2 of body area
  5 minutes post induction | -0.4 (0.4) | -0.3 (0.4)
  10 minutes post induction | -0.6 (0.6) | -0.5 (0.5)
Statistical Analysis 1: Comparison: Propofol vs Ketofol; Average change in Cardiac Index (CI) from baseline to 5 minutes post induction was compared between treatment groups; Test type: Superiority or Other; p = 0.26, t-test, 2 sided; Mean Difference (Final Values) = 0.1, 95% CI 2-sided [-0.1 to 0.3]
Statistical Analysis 2: Comparison: Propofol vs Ketofol; Average change in Cardiac Index (CI) from baseline to 10 minutes post induction was compared between treatment groups; Test type: Superiority or Other; p = 0.71, t-test, 2 sided; Mean Difference (Final Values) = 0.0, 95% CI 2-sided [-0.2 to 0.3]

6. Secondary Outcome: Average Change in Heart Rate (HR)
Description: HR was recorded every minute for a total of 30 minutes after anesthesia was induced and readings were captured via a Non-Invasive Cardiac Output Monitor [NICOM], Cheetah Medical, Israel. The average change in HR (as compared to baseline HR) during the specified time intervals is reported.
Time Frame: Baseline, 5 minutes, 10 minutes post induction
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Propofol | Ketofol
Number analyzed (Participants) | 43 | 41
Beats per minute
  5 minutes post induction | -4.0 (4.5) | -4.6 (6.0)
  10 minutes post induction | -5.2 (5.2) | -7.0 (8.0)
Statistical Analysis 1: Comparison: Propofol vs Ketofol; Average heart rate from baseline to 5 minutes post induction was compared between treatment groups; Test type: Superiority or Other; p = 0.61, t-test, 2 sided; Mean Difference (Final Values) = -0.6, 95% CI 2-sided [-2.9 to 1.7]
Statistical Analysis 2: Comparison: Propofol vs Ketofol; Average heart rate from baseline to 10 minutes post induction was compared between treatment groups; Test type: Superiority or Other; p = 0.22, t-test, 2 sided; Mean Difference (Final Values) = -1.8, 95% CI 2-sided [-4.8 to 1.1]

7. Secondary Outcome: Average Change in Systolic Blood Pressure (SBP)
Description: Blood pressure was recorded every minute for a total of 30 minutes after anesthesia was induced and readings were captured via a Non-Invasive Cardiac Output Monitor [NICOM], Cheetah Medical, Israel. The average change in SBP (as compared to baseline SBP) during the specified time intervals is reported.
Time Frame: Baseline, 5 minutes, 10 minutes post induction
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Propofol | Ketofol
Number analyzed (Participants) | 43 | 41
mmHg
  5 minutes post induction | -26.3 (16.2) | -12.5 (12.4)
  10 minutes post induction | -30.6 (16.6) | -21.8 (16.8)
Statistical Analysis 1: Comparison: Propofol vs Ketofol; Average change in Systolic Blood Pressure from baseline to 5 minutes post induction was compared between treatment groups; Test type: Superiority or Other; p < 0.001, t-test, 2 sided; Mean Difference (Final Values) = 13.7, 95% CI 2-sided [7.5 to 20.0]
Statistical Analysis 2: Comparison: Propofol vs Ketofol; Average change in Systolic Blood Pressure from baseline to 10 minutes post induction was compared between treatment groups; Test type: Superiority or Other; p = 0.017, t-test, 2 sided; Mean Difference (Final Values) = 8.8, 95% CI 2-sided [0.2 to 9.5]

8. Secondary Outcome: Average Change in Diastolic Blood Pressure (DBP)
Description: Blood pressure was recorded every minute for a total of 30 minutes after anesthesia was induced and readings were captured via a Non-Invasive Cardiac Output Monitor [NICOM], Cheetah Medical, Israel. The average change in DBP (as compared to baseline DBP) during the specified time intervals is reported.
Time Frame: Baseline, 5 minutes, 10 minutes post induction
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Propofol | Ketofol
Number analyzed (Participants) | 43 | 41
mmHg
  5 minutes post induction | -15.9 (11.3) | -8.8 (9.1)
  10 minutes post induction | -19.3 (11.5) | -14.5 (9.8)
Statistical Analysis 1: Comparison: Propofol vs Ketofol; Average change in Diastolic Blood Pressure from baseline to 5 minutes post induction was compared between treatment groups; Test type: Superiority or Other; p < 0.01, t-test, 2 sided; Mean Difference (Final Values) = 7.1, 95% CI 2-sided [2.7 to 11.5]
Statistical Analysis 2: Comparison: Propofol vs Ketofol; Average change in Diastolic Blood Pressure from baseline to 10 minutes post induction was compared between treatment groups; Test type: Superiority or Other; p = 0.042, t-test, 2 sided; Mean Difference (Final Values) = 4.8, 95% CI 2-sided [0.2 to 9.5]

9. Secondary Outcome: Average Change in Mean Arterial Pressure (MAP)
Description: MAP was recorded every minute for a total of 30 minutes after anesthesia was induced and readings were captured via a Non-Invasive Cardiac Output Monitor [NICOM], Cheetah Medical, Israel. The average change in MAP from baseline during the specified time intervals is reported.
  MAP is a term used in medicine to describe an average blood pressure in an individual. It is defined as the average arterial pressure during a single cardiac cycle.
Time Frame: Baseline, 5 minutes, 10 minutes post induction
Population: The analysis population of 43/40 (vs. 43/41 at baseline) is due to the NICOM not functioning properly during certain aspects of the procedure and therefore, did not provide a number.
Measure: Mean (Standard Deviation); unit: Millimeters of mercury (mmHg)
Arm/Group | Propofol | Ketofol
Number analyzed (Participants) | 43 | 40
Millimeters of mercury (mmHg)
  5 minutes post induction | -18.7 (11.5) | -9.3 (9.4)
  10 minutes post induction | -22.6 (11.7) | -16.2 (11.1)
Statistical Analysis 1: Comparison: Propofol vs Ketofol; Average change in Mean Arterial Pressure (MAP) from baseline to 5 minutes post induction was compared between treatment groups; Test type: Superiority or Other; p < 0.001, t-test, 2 sided; Mean Difference (Final Values) = 9.4, 95% CI 2-sided [4.8 to 13.9]
Statistical Analysis 2: Comparison: Propofol vs Ketofol; Average change in Mean Arterial Pressure from baseline to 10 minutes post induction was compared between treatment groups; Test type: Superiority or Other; p = 0.013, t-test, 2 sided; Mean Difference (Final Values) = 6.3, 95% CI 2-sided [1.4 to 11.3]

10. Secondary Outcome: Average Change in Total Peripheral Resistance (TPR)
Description: TPR was recorded every minute for a total of 30 minutes after anesthesia was induced and readings were captured via a Non-Invasive Cardiac Output Monitor [NICOM], Cheetah Medical, Israel. The average change in TPR from baseline during the specified time intervals is reported. TPR is the overall resistance to blood flow through the systemic blood vessels.
Time Frame: Baseline, 5 minutes, 10 minutes post induction
Population: The analysis population of 39/38 (vs. 43/41 at baseline) is due to the NICOM not functioning properly during certain aspects of the procedure and therefore, did not provide a number.
Measure: Mean (Standard Deviation); unit: dynes * sec/cm^-5
Arm/Group | Propofol | Ketofol
Number analyzed (Participants) | 39 | 38
dynes * sec/cm^-5
  5 minutes post induction | -261.2 (211.9) | -147.6 (161.8)
  10 minutes post induction | -321.7 (251.3) | -235.0 (226.5)
Statistical Analysis 1: Comparison: Propofol vs Ketofol; Average change in Total Peripheral Resistance (TPR) from baseline to 5 minutes post induction was compared between treatment groups; Test type: Superiority or Other; p < 0.01, t-test, 2 sided; Mean Difference (Final Values) = 113.6, 95% CI 2-sided [28.1 to 199.1]
Statistical Analysis 2: Comparison: Propofol vs Ketofol; Average change in Total Peripheral Resistance (TPR) from baseline to 10 minutes post induction was compared between treatment groups; Test type: Superiority or Other; p = 0.12, t-test, 2 sided; Mean Difference (Final Values) = 86.8, 95% CI 2-sided [-21.7 to 195.3]

11. Secondary Outcome: Average Change in Total Peripheral Resistance Index (TPRI)
Description: TPRI was recorded every minute for a total of 30 minutes after anesthesia was induced and results were captured via a Non-Invasive Cardiac Output Monitor [NICOM], Cheetah Medical, Israel. The average change in TPRI from baseline during the specified time intervals is reported.
Time Frame: Baseline, 5 minutes, 10 minutes post induction
Population: The analysis population of 39/39 (vs. 43/41 at baseline) is due to the NICOM not functioning properly during certain aspects of the procedure and therefore, did not provide a number.
Measure: Mean (Standard Deviation); unit: dynes * sec/cm^-5/m^2
Arm/Group | Propofol | Ketofol
Number analyzed (Participants) | 39 | 39
dynes * sec/cm^-5/m^2
  5 minutes post induction | -457.6 (362.4) | -275.0 (293.2)
  10 minutes post induction | -559.3 (421.0) | -430.6 (407.5)
Statistical Analysis 1: Comparison: Propofol; Average change in Total Peripheral Resistance Index (TPRI) from baseline to 5 minutes post induction was compared between treatment groups; Test type: Superiority or Other; p = 0.017, t-test, 2 sided; Mean Difference (Final Values) = 182.6, 95% CI 2-sided [33.8 to 331.3]
Statistical Analysis 2: Comparison: Propofol vs Ketofol; Average change in Total Peripheral Resistance Index (TPRI) from baseline to 10 minutes post induction was compared between treatment groups; Test type: Superiority or Other; p = 0.17, t-test, 2 sided; Mean Difference (Final Values) = 128.7, 95% CI 2-sided [-58.1 to 315.5]

12. Secondary Outcome: Average Change in Stroke Volume (SV)
Description: SV was recorded every minute for a total of 30 minutes after anesthesia was induced and results were captured via a Non-Invasive Cardiac Output Monitor [NICOM], Cheetah Medical, Israel. The average change in SV from baseline during the specified time intervals is reported. SV is the milliliters of blood ejected during each contraction of the heart.
Time Frame: Baseline, 5 minutes, 10 minutes post induction
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Milliliters of blood per beat
Arm/Group | Propofol | Ketofol
Number analyzed (Participants) | 41 | 40
Milliliters of blood per beat
  5 minutes post induction | -12.2 (10) | -7.8 (7.8)
  10 minutes post induction | -16.4 (12.8) | -11.6 (8.7)
Statistical Analysis 1: Comparison: Propofol vs Ketofol; Average change in Stroke Volume (SV) from baseline to 5 minutes post induction was compared between treatment groups; Test type: Superiority or Other; p = 0.029, t-test, 2 sided; Mean Difference (Final Values) = 4.4, 95% CI 2-sided [0.5 to 8.4]
Statistical Analysis 2: Comparison: Propofol vs Ketofol; Average change in Cardiac Index (CI) from baseline to 10 minutes post induction was compared between treatment groups; Test type: Superiority or Other; p = 0.051, t-test, 2 sided; Mean Difference (Final Values) = 4.8, 95% CI 2-sided [-0.0 to 9.7]

13. Secondary Outcome: Average Change in Stroke Volume Index (SVI)
Description: SVI was recorded every minute for a total of 30 minutes after anesthesia was induced and results were captured via a Non-Invasive Cardiac Output Monitor [NICOM], Cheetah Medical, Israel. The average change in SVI (as compared to baseline SVI) during the specified time intervals is reported. To determine SVI, stroke volume is divided by the body surface area in order to account for body size.
Time Frame: Baseline, 5 minutes, 10 minutes post induction
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Milliters per beat per m^2 of body area
Arm/Group | Propofol | Ketofol
Number analyzed (Participants) | 41 | 40
Milliters per beat per m^2 of body area
  5 minutes post induction | -6.8 (5.6) | -4.3 (4.3)
  10 minutes post induction | -9.2 (6.8) | -6.6 (4.9)
Statistical Analysis 1: Comparison: Propofol vs Ketofol; Average change in Stroke Volume Index (SVI) from baseline to 5 minutes post induction was compared between treatment groups; Test type: Superiority or Other; p = 0.027, t-test, 2 sided; Mean Difference (Final Values) = 2.5, 95% CI 2-sided [0.3 to 4.7]
Statistical Analysis 2: Comparison: Propofol vs Ketofol; Average change in Stroke Volume Index (SVI) from baseline to 10 minutes post induction was compared between treatment groups; Test type: Superiority or Other; p = 0.052, t-test, 2 sided; Mean Difference (Final Values) = 2.6, 95% CI 2-sided [-0.0 to 5.2]

14. Secondary Outcome: Average Change in Stroke Volume Variation (SVV)
Description: SVV was recorded every minute for a total of 30 minutes after anesthesia was induced and results were captured via a Non-Invasive Cardiac Output Monitor [NICOM], Cheetah Medical, Israel. SVV is a dynamic flow-based parameter and together with cardiac output provides an indication of fluid responsiveness. The average change in SVV (as compared to baseline SVV) during the specified time intervals is reported. SVV is calculated by taking the SVmax - SVmin /*100/ SV mean.
Time Frame: Baseline, 5 minutes, 10 minutes post induction
Population: The analysis population of 38/35 (vs. 43/41 at baseline) is due to the NICOM not functioning properly during certain aspects of the procedure and therefore, did not provide a number.
Measure: Mean (Standard Deviation); unit: Percentage of mean stroke volume
Arm/Group | Propofol | Ketofol
Number analyzed (Participants) | 38 | 35
Percentage of mean stroke volume
  5 minutes post induction | -2.2 (2.0) | -2.6 (2.2)
  10 minutes post induction | -2.6 (2.1) | -3.1 (2.4)
Statistical Analysis 1: Comparison: Propofol vs Ketofol; Average change in Stroke Volume Variation (SVV) from baseline to 5 minutes post induction was compared between treatment groups; Test type: Superiority or Other; p = 0.44, t-test, 2 sided; Mean Difference (Final Values) = -0.4, 95% CI 2-sided [-1.4 to 0.6]
Statistical Analysis 2: Comparison: Propofol vs Ketofol; Average change in Stroke Volume Variation (SVV) from baseline to 10 minutes post induction was compared between treatment groups; Test type: Superiority or Other; p = 0.37, t-test, 2 sided; Mean Difference (Final Values) = -0.5, 95% CI 2-sided [-1.6 to 0.6]

ADVERSE EVENTS:
Time Frame: Baseline to 30 minutes post induction of anesthesia
Arm/Group | Propofol | Ketofol
Serious Adverse Events (participants affected / at risk) | 0/43 | 0/42
Other Adverse Events (participants affected / at risk) | 0/43 | 0/42

LIMITATIONS AND CAVEATS:
The dose ratio implemented was not ideal. Enrollment was limited to ASA I and II patients only.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No